CLINICAL TRIAL: NCT00437346
Title: Study of Gastroscopy Negative Dyspepsia - Effect of Acid-reducing Treatment and Information on Various Types of Dysmotility.
Brief Title: Functional Dyspepsia - Effect of Acid-Reducing Treatment and Information.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The project leader left our hospital and the project were shut down.
Sponsor: Helse Fonna (Other)
Responsible Party: Principal Investigator, Helge Børresen, Dr., Helse Fonna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15312
Record Dates: First submitted 2007-02-15; First posted 2007-02-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Dyspepsia
Keywords: dyspepsia; functional dyspepsia; treatment; drug therapy; information
MeSH Terms: conditions — Dyspepsia

ARMS (2):
- Group A (Active Comparator): Patients is given thorough information based on the tests taken plus medical treatment.
  Interventions: Procedure: Individualized and comprehensive information; Drug: Lanzo Melt
- Group B (Active Comparator): Patients receive simple written information based on the tests taken plus medical treatment.
  Interventions: Drug: Lanzo Melt

INTERVENTIONS:
Procedure: Individualized and comprehensive information — Thorough verbal and written information about results of the tests. Individualized meals recommendation based on the results.
  Arms: Group A
Drug: Lanzo Melt — 30mg, od, 1/2 h before meal
  Arms: Group A
Drug: Lanzo Melt — 30mg, od, 1/2 h before meal
  Arms: Group B

SUMMARY:
Study title: Functional dyspepsia -- effect of acid reducing treatment and individualized information.

Summary: 15-20% of all people experience dyspepsia each year. Dyspepsia means pain or discomfort in the upper part of the abdomen. Accompanying symptoms from the esophagus may be present. The most important relevant medical examination is gastroscopy, and if the findings are normal the condition is usually classified as functional dyspepsia.

Several disturbances of function are now known as potential causes of such symptoms, and the optimal choice of treatment may vary.

In the study the investigators plan to examine whether different types of functional disturbances respond differently to medical therapy. In particular, the investigators want to assess whether comprehensive and individualized information will influence the results of therapy. This has not been previously studied systematically.

The investigators also postulate that disturbances of function of the esophagus may cause complaints that should be classified as functional dyspepsia even if the symptoms are atypical. Few studies have been done to evaluate this hypothesis, and there may be potential consequences for choice of appropriate treatment.

In animal models and in humans is recently demonstrated that elevated gastric pH because of anti-ulcer treatment can trigger food allergy. We use a proton pump inhibitor in our study and eventually development of food allergy will influence patient's condition in an observations period. That why we're observing IgE dynamics in our study.

DETAILED DESCRIPTION:
Purpose

Functional dyspepsia is a common disorder affecting approximately 25 % of the adult population. Functional dyspepsia is defined from symptoms according to the Rome II criteria. A normal upper endoscopy is also warranted Many of these patients have specific motility disorders. A more accurate diagnosis could mean a more effective treatment.

In this study the patients take several tests in order to make a more specific diagnosis. These include: 24 hour pH-monitoring, oesophagusmanometry, drink test and scintigrafy.

We will study the effect of acid reducing treatment (proton pump inhibitors) on the different dysmotility-types and also the effect of medical information and advise.

We will observe concentrations of total IgE and various specific antibodies against food allergens in serum when taking PPI. Results here can vary dependent on whether the patient has used PPI anytime before or not.

Patients

The patients are included via referrals from general practitioners and hospital doctors. An upper endoscopy is performed. If this investigation is normal the patient is considered for inclusion in the study.

Criteria for inclusion are

* Age 20 - 60 years
* Rome II criteria fulfilled
* Helicobacter test negative (urease-test)
* Informed consent

Criteria for exclusion are

* Diabetes
* Prior gastrointestinal surgery
* Treatment with proton pump inhibitors / H2 blockers the last 30 days
* Pregnancy / lactation
* Current use of NSAIDs
* Serious psychiatric illness
* Serious egg-allergy

Study design

Start of the study: symptom score based on symptoms within the last three days. Lanzo melt 30 mg daily is given as a morning dose. Patients are randomized in two groups. Group A is given thorough information based on the tests taken plus medical treatment. Group B receives medical treatment only.

After two weeks symptom score per telephone. After four weeks a new symptom score. A reduction by at least 25 % is defined as treatment response. These patients continue their medical treatment for three months. Now all patients receive thorough information.

Non responders end their medical treatment and they are followed with medical information and advise the next three months.

After eight weeks symptom score per telephone. After 12 weeks symptom score per telephone. After 16 weeks the study is ended. Symptom score is taken.

After 4 and 16 weeks the patient evaluates his/her treatment in five categories: Very satisfied, satisfied, less satisfied, no change, worse.

Symptom score

Seven symptoms are scored from 1-7 points based on the last week. The symptoms are: regurgitation, nausea, early satiety, belching, pain referred to meals, pain not referred to meals, postprandial fullness.

1. No symptoms
2. Insignificant symptoms (as usual ignored)
3. Light symptoms (easy to ignore)
4. Moderate symptoms (easy to tolerate)
5. Quite marked symptoms (not easy to tolerate)
6. Marked symptoms (affects daily activities)
7. Substantional symptoms (can't do daily activities)

24 hour pH monitoring

Digitrapper III from Synectics is used. A probe is installed trans nasally to the gastric lumen where a pH value is registered. Afterwards the probe is placed five cm over the upper border of the lower esophageal sphincter (LES). After 24 hours registration is completed and analyzed with the use of Polygram 98 from Medtronic Functional Diagnostics AS.

Total reflux index, reflux with meals, postprandial reflux, nightly reflux and long reflux episodes are registered. Pathologic reflux index is defined as pathological if reflux is over 5 %.

Acid Clearence Time (ACT) is also estimated. It is found by dividing total reflux time with the number of refluxes. Upper normal limit is set to 0,85 minutes/reflux.

Esophagusmanometry

We use perfusion manometry. The catheter has sensors in five levels five cm apart. LES is first localized and length and resting pressure are registered. We test for normal relaxation with swallowing. Then we test the motility (peristalsis and amplitude/duration of pressure waves).

Scintigraphy

We give a standard meal composed of two omelets, one slice of bread and a glass of water. Radioactive Technesium is injected into the omelet and the meal is eaten in ten minutes. Picture uptakes are taken according to the protocol the first hour after completion of the meal. Gastric emptying time is estimated.

Drink test The patients drink water 150 ml/min until they feel they must stop. Symptoms are registered when they stop and 15 and 30 minutes there after. This is a test to determine accommodation and visceral sensibility.

Blood tests Hemoglobin, sedimentation rate, CRP, leucocytes, thrombocytes, bilirubin, ALP, ALAT, g-GT, albumin and amylase are taken to exclude organic disease. It does not represent a variable in the study design.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 60 years
* Rome II criteria fulfilled
* Helicobacter test negative (urease-test)
* Informed consent

Exclusion Criteria:

* Diabetes
* Prior gastrointestinal surgery
* Treatment with proton pump inhibitors / H2 blockers the last 30 days
* Pregnancy / lactation
* Current use of NSAIDs
* Serious psychiatric illness
* Serious egg allergy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Improvement of symptom score | november 2009-2013

CONTACTS AND LOCATIONS:
Overall Officials: Valerij Glazkov, MD, Principal Investigator — Department of Medicine, Haugesund Hospital, N-5504 Haugesund, Norway; Jan G. Hatlebakk, MD, PhD, Study Chair — Department of Medicine, Haukeland University Hospital, 5021 Bergen, Norway
Locations (5):
- Norway (5):
  - Department of Medicine, Haugesund Hospital, Haugesund
  - Department of Medisin, Haugesund Hospital, Haugesund
  - Department of Radiology, Haugesund Hospital, Haugesund
  - Surgical Department, Haugesund Hospital, Haugesund
  - Gastro-group, Haugesund

REFERENCES:
- [Background] Talley NJ, Stanghellini V, Heading RC, Koch KL, Malagelada JR, Tytgat GN. Functional gastroduodenal disorders. Gut. 1999 Sep;45 Suppl 2(Suppl 2):II37-42. doi: 10.1136/gut.45.2008.ii37. PMID 10457043
- [Background] Tack J, Bisschops R, Sarnelli G. Pathophysiology and treatment of functional dyspepsia. Gastroenterology. 2004 Oct;127(4):1239-55. doi: 10.1053/j.gastro.2004.05.030. No abstract available. PMID 15481001
- [Background] Talley NJ, Verlinden M, Jones M. Can symptoms discriminate among those with delayed or normal gastric emptying in dysmotility-like dyspepsia? Am J Gastroenterol. 2001 May;96(5):1422-8. doi: 10.1111/j.1572-0241.2001.03683.x. PMID 11374677
- [Background] Talley NJ, Locke GR, Lahr BD, Zinsmeister AR, Cohard-Radice M, D'Elia TV, Tack J, Earnest DL. Predictors of the placebo response in functional dyspepsia. Aliment Pharmacol Ther. 2006 Apr 1;23(7):923-36. doi: 10.1111/j.1365-2036.2006.02845.x. PMID 16573795
- [Background] Bolling-Sternevald E, Lauritsen K, Aalykke C, Havelund T, Knudsen T, Unge P, Ekstrom P, Jaup B, Norrby A, Stubberod A, Melen K, Carlsson R, Jerndal P, Junghard O, Glise H. Effect of profound acid suppression in functional dyspepsia: a double-blind, randomized, placebo-controlled trial. Scand J Gastroenterol. 2002 Dec;37(12):1395-402. doi: 10.1080/003655202762671260. PMID 12523588
- [Background] Talley NJ, Vakil N; Practice Parameters Committee of the American College of Gastroenterology. Guidelines for the management of dyspepsia. Am J Gastroenterol. 2005 Oct;100(10):2324-37. doi: 10.1111/j.1572-0241.2005.00225.x. PMID 16181387
- [Background] Jones MP, Roth LM, Crowell MD. Symptom reporting by functional dyspeptics during the water load test. Am J Gastroenterol. 2005 Jun;100(6):1334-9. doi: 10.1111/j.1572-0241.2005.40802.x. PMID 15929766
- [Background] Untersmayr E, Jensen-Jarolim E. The effect of gastric digestion on food allergy. Curr Opin Allergy Clin Immunol. 2006 Jun;6(3):214-9. doi: 10.1097/01.all.0000225163.06016.93. PMID 16670517